CLINICAL TRIAL: NCT00375193
Title: A Phase 2 Trial of Single-Agent Amrubicin in Patients With Extensive Disease Small Cell Lung Cancer That is Refractory or Progressive Within 90 Days of Completion of First Line Platinum-based Chemotherapy
Brief Title: Study of Amrubicin in Patients With Small Cell Lung Cancer Refractory or Progressive to Prior Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNF3140-SCLC-002
Record Dates: First submitted 2006-09-09; First posted 2006-09-12 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Small Cell Lung Cancer
Keywords: small cell lung cancer; amrubicin
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — amrubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Amrubicin 40mg/m<2> IV days 1, 2, 3 of each 21-day cycle until cycle 6 or no longer beneficial.
  Interventions: Drug: Amrubicin

INTERVENTIONS:
Drug: Amrubicin — Amrubicin 40mg/m<2> IV days 1, 2, 3 of each 21-day cycle until Cycle 6 or no longer beneficial

SUMMARY:
The purpose of the study is to evaluate the objective tumor response rate of amrubicin when administered as second-line therapy to ED-SCLC patients who have refractory or progressive disease.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of SCLC; extensive-disease (ED) at time of study entry
* Refractory to first-line platinum-based chemotherapy (i.e., has received one prior platinum-based chemotherapy regimen) defined as one of the following:

  * Best response to first-line chemotherapy is radiographically documented progression (refractory disease)
  * Best response to first-line chemotherapy is radiographically documented response or stable disease, with subsequent documented progression during continuing chemotherapy (resistant relapse)
  * Documented progression within 90 days of completion of first-line chemotherapy (last dose of chemotherapy), regardless of best response to treatment (resistant relapse)
* At least 18 years of age
* ECOG Performance Status of 0, 1, or 2
* Measurable disease defined by RECIST criteria

  * Measurable disease: The presence of at least one measurable lesion. If only one lesion is present, the neoplastic nature of the disease site should be confirmed by histology and/or cytology.
  * Measurable lesion: Lesions that can be accurately measured in at least one dimension with the longest diameter ≥20mm using conventional techniques or ≥10mm using spiral CT scans.
* CT (including spiral CT) scans and MRI are the preferred methods of measurement; however, chest x-rays are acceptable if the lesions are clearly defined and surrounded by aerated lung. Clinically detected lesions will only be considered measurable when they are superficial (e.g., skin nodules and palpable lymph nodes). For the case of skin lesions, documentation by color photography, including a ruler to estimate the size of the lesion is required.
* Adequate organ function including the following:

  * Adequate bone marrow reserve: absolute neutrophil (segmented and bands) count (ANC) ≥1500 cells/μL, platelet count ≥100,000 cells/μL and hemoglobin ≥9g/dL.
  * Hepatic: bilirubin ≤ 1.5 X ULN; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 X ULN.
  * Renal: serum creatinine < 2.0 mg/dL or calculated creatinine clearance >60 mL/min.
  * Cardiac: Left ventricular ejection fraction (LVEF) ≥ 50% by MUGA or echocardiography (intra-patient reassessment of LVEF should be performed via the same method throughout the study).
* Negative serum pregnancy test at the time of enrollment for women of child-bearing potential. For men and women of child-bearing potential, use of effective contraceptive methods during the study.
* Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and to return for the required assessments.

Exclusion Criteria:

* Pregnant or nursing women
* Chest radiotherapy within the previous 28 days or other radiotherapy within the previous 14 days. Recovery from the acute toxic effects of radiation required prior to study enrollment. Measurable lesions that have been previously irradiated must be enlarging to be considered target lesions. Prior radiation therapy allowed to < 25% of the bone marrow.
* More than 1 prior chemotherapy regiment for SCLC
* Prior anthracycline treatment
* Treatment with any investigational agent within 28 days or standard chemotherapy within 21 days prior to first dose. Patients must have recovered from all acute adverse effecxts of prior therapies, excluding alopecia
* Patients with secondary primary malignancy (except in situ carcinoma of the cervix or adequately treated nonmelanomatous carcinoma of the skin or other malignancy treated at least 2 years previously with surgery and/or radiotherapy and no evidence of recurrence since that time)
* Concurrent severe or uncontrolled medical disease (i.e., active systemic infection, diabetes, hypertension, coronary artery disease, congestive heart failure) that, in the opinion of the Investigator, would compromise the safety of the patient or compromise the ability of the patient to complete the study.
* Symptomatic central nervous system metastases. Patients with asymptomatic brain metastases are allowed. The patient must be stable after radiotherapy for ≥ 2 weeks and off corticosteroids for ≥ 1 week.
* History of interstitial lung disease or pulmonary fibrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2006-11-01 (Actual); Primary Completion 2008-05-01 (Actual); Study Completion 2009-03-01 (Actual)

PRIMARY OUTCOMES:
Objective tumor response rate according to RECIST | Until Disease Progression

SECONDARY OUTCOMES:
Duration of overall response | Until Disease Progression
Time to tumor progression | Until Disease Progression
Progression free survival | Until death or disease progression
Overall survival | Until death
Toxicity profile | Until 30 days after final dose
Incidence of cardiomyopathy | Until end of study participation
Incidence of CNS progression | Until disease progression
Pharmacokinetic parameters | Cycle 1 only

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Ungerleider, MD, Study Director — Theradex
Locations (46):
- United States (44):
  - Hematology Oncology Associates, Phoenix, Arizona
  - Rocky Mountain Cancer Center - Sky Ridge, Lone Tree, Colorado
  - Ocala Oncology Center, Ocala, Florida
  - Cancer Centers of Florida, PA, Ocoee, Florida
  - John B. Amos Cancer Center, Columbus, Georgia
  - Cancer Care & Hematology Specialists of Chicago, Niles, Illinois
  - Oncology & Hematology of Central Illinois, Peoria, Illinois
  - Blessing Cancer Center, Quincy, Illinois
  - Central Indiana Cancer Centers - Indianapolis, Indianapolis, Indiana
  - Norton Healthcare - Louisville Oncology, Louisville, Kentucky
  - Maryland Oncology Hematology, PA, Columbia, Maryland
  - Alliance Hematology Oncology, PA - Carroll County Cancer Center, Westminster, Maryland
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Minnesota Onc/Hem, PA - Minneapolis, Minneapolis, Minnesota
  - University of MN/Division of Hematology, Oncology & Transplantation, Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - St. Joseph Oncology, Inc., Saint Joseph, Missouri
  - Arch Medical Group - Arch Medical Services, Inc., St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New York Oncology Hematology, PC, Albany, New York
  - SUNY Upstate Medical Center, Syracuse, New York
  - Northwestern Carolina Oncology & Hematology, Hickory, North Carolina
  - Raleigh Hematology Oncology Associates, Raleigh, North Carolina
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Medical Oncology Associates, Kingston, Pennsylvania
  - University of Tennessee Medical Center, Knoxville, Knoxville, Tennessee
  - Sarah Cannon, Nashville, Tennessee
  - Texas Oncology - Amarillo, Amarillo, Texas
  - Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Oncology, PA - Bedford, Bedford, Texas
  - Texas Cancer Center at Medical City, Dallas, Texas
  - Texas Oncology, P.A. - Dallas, Dallas, Texas
  - Texas Oncology, P.A., Sammons Cancer Center, Dallas, Texas
  - Texas Oncology, PA - Fort Worth, Fort Worth, Texas
  - West Texas Cancer Center, Odessa, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texas Oncology Cancer Care and Research Center, Waco, Texas
  - Texas Oncology, PA - Deke Slayton Cancer Center, Webster, Texas
  - Texas Oncology - Wichita Falls, Wichita Falls, Texas
  - Virginia Oncology Associates - Norfolk, VA, Norfolk, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Inc., Salem, Virginia
  - Puget Sound Cancer Center, Seattle, Washington
  - Northwest Cancer Specialists - Vancouver Cancer Center, Vancouver, Washington
  - Yakima Regional Cancer Care Center - North Star Lodge Cancer Center, Yakima, Washington
- Free University Medical Center, Amsterdam, Netherlands
- Royal Marsden Hospital in Downs Road, Sutton, Surrey, United Kingdom

REFERENCES:
- [Background] Ettinger DS, Jotte R, Lorigan P, Gupta V, Garbo L, Alemany C, Conkling P, Spigel DR, Dudek AZ, Shah C, Salgia R, McNally R, Renschler MF, Oliver JW. Phase II study of amrubicin as second-line therapy in patients with platinum-refractory small-cell lung cancer. J Clin Oncol. 2010 May 20;28(15):2598-603. doi: 10.1200/JCO.2009.26.7682. Epub 2010 Apr 12. PMID 20385980
- [Background] Spigel DR, et al. Amrubicin (AMR) and cardiotoxicity in second-line treatment of small cell lung cancer (SCLC): A pooled analysis of left ventricular ejection fraction (LVEF) in two phase II trials. 2009 ASCO Annual Meeting, May 29-June 2, 2009, Chicago, IL. Abstract No.e19019. J Clin Oncol 2009;27(suppl)